CLINICAL TRIAL: NCT05892042
Title: Assessment of Anti-Coagulation Therapy on Patient With Left Ventricular Thrombus After ST Segment Elevation Myocardial Infarction
Brief Title: Anti-CoagulaTion on Left Ventricular Thrombus After ST Segment Elevation Myocardial Infarction
Acronym: ACTonLVT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jilin University (Other)
Responsible Party: Principal Investigator, Mingyou Zhang, Associate prof, Jilin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACT on LVT
Record Dates: First submitted 2023-05-28; First posted 2023-06-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-05

CONDITIONS: ST-segment Elevation Myocardial Infarction (STEMI); Left Ventricular Thrombus
Keywords: STEMI, LVT, Anticoagulation
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Rivaroxaban

STUDY DESIGN:
Intervention Model Description: Acute ST segment elevation myocardial infarction complicated with left ventricular thrombus weather or not treated with primary PCI.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention (Experimental): patient will receive dual antiplatelet therapy, the choose of p2Y12 inhibitor is at the discretion of the clinician. in addition the patient will receive rivaroxaban 15mg daily in addition to the dual antiplatelet therapy.
  Interventions: Drug: Rivaroxaban 15 MG [Xarelto]
- control (No Intervention): patient will receive dual antiplatelet therapy, the choose of p2Y12 inhibitor is at the discretion of the clinician.

INTERVENTIONS:
Drug: Rivaroxaban 15 MG [Xarelto] — Eligible subjects randomized into experimental group will receive rivaroxaban 15mg daily in addition to dual anti platelet therapy unless confirmed resolution of the left ventricular thrombus.
  Other Names: Xarelto
  Arms: intervention

SUMMARY:
Contemporary data are lacking regarding the management of left ventricular thrombus (LVT) developed after ST segment elevation myocardial infarction

DETAILED DESCRIPTION:
Left ventricular thrombus (LVT) is a commom complication after ST segment elevation myocardial infarction (STEMI), reperfusion therapy have reduced the incidence of LVT, however, about 6% of all STEMI patients will develop LVT. the risk of LVT development in anterior STEMI with reduced LVEF are as high as 20%. Although current guideline recommend anti-coagulation therapy, but the evidence still based on observational data, there has been inconsistency with the benefit of the coagulation therapy, give the significant increased bleeding risk by superimpose anti-coagulation therapy to the dual anti-platelet therapy. especially in the era of more potent anti-platelet P2Y12 inhibitor widely used clinical. the mechanism of LVT is different from that of the atrial fibrillation in which the risk of systemic embolism is persistent, coagulation bring absolute clinical benefit for high risk patients. however, for LVT developed following STEMI tend to be temporary, majority of thrombus resolve within 1-3 months after STEMI event. more likely a reflection of coagulation system in response to the necrosis of infarct myocardium. The optimal management in LVT after STEMI warrants further exploration. the desiring of randomized controlled clinical trial to compare dual anti platelet + anti-coagulation and dual anti-platelet without anti-coagulation in patient LVT are justified.

ELIGIBILITY:
Inclusion Criteria:

Established ST segment elevation myocardial infarction within 7 days Left ventricular thrombus (LVT) is detected by either cardiac magnetic resonance (CMR) or TTE.

Ongoing treatment with dual anti-platelet therapy according to ESC/AHA guidelines at the time of randomization

Exclusion Criteria:

Clinically or hemodynamically unstable planed major surgeon such as CABG or Valve replacement within next 12 months Concomitant condition that requires anti- coagulation therapy, such as AF, DVT.

Any contraindication of anticoagulant therapy History of intracranial hemorrhage; Woman who is currently pregnant, or breastfeeding serious impaired renal and liver functions life expectancy less than 1 year can not provide consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with the first occurrence of Stroke and other systemic embolism | 12 months
  The percentage of participants with the first occurrence of Stroke and other systemic embolism were evaluated.

SECONDARY OUTCOMES:
Composite major adverse events | 12 months
  The incidence of a composite adverse events, including all cause mortality, recurrent myocardial infarction, ischemic stroke and other systemic embolism
LVT resolution | 12 months
  the LVT resolve will be determined monthly by follow-up imaging examination (Echo cardiograph or Cardiac magnetic resonance). The percentage of LVT resolve at 3 months will be calculated for each group.
Total LVT present time | 12 months
  LVT will be followed every month in the first 3 months, every 3 months thereafter to determine the present of LVT by Echo cardiograph or Cardiac magnetic resonance.
Percentage of Participants With Clinically Significant Bleeding | 12 months
  Clinically significant bleeding is a composite of Thrombolysis in Myocardial Infarction (TIMI) major bleeding, minor bleeding, and bleeding requiring medical attention (BRMA). TIMI major bleeding is defined as any symptomatic intracranial hemorrhage, clinically overt signs of hemorrhage (including imaging) associated with a drop in hemoglobin of greater than or equal to (>=) 5 grams per deciliter (g/dL) (or when the hemoglobin concentration is not available, an absolute drop in hematocrit of >=15 percent (%)). TIMI minor bleeding event is defined as any clinically overt sign of hemorrhage (including imaging) that is associated with a fall in hemoglobin concentration of 3 to less than (<) 5 g/dL (or, when hemoglobin concentration is not available, a fall in hematocrit of 9 percent to <15 percent). A BRMA event is defined as any bleeding event that requires medical treatment, surgical treatment, or laboratory evaluation, and does not meet criteria for a major or minor bleeding event.
Percentage of Participants With Thrombolysis in Myocardial Infarction (TIMI) Major Bleeding | 12 months
  TIMI major bleeding is defined as any symptomatic intracranial hemorrhage, Clinically overt signs of hemorrhage (including imaging) associated with a drop in hemoglobin of >= 5 g/dL (or when the hemoglobin concentration is not available, an absolute drop in hematocrit of >=15 percent
Percentage of Participants With Thrombolysis in Myocardial Infarction (TIMI) Minor Bleeding | 12 months
  TIMI minor bleeding event is defined as any clinically overt sign of hemorrhage (including imaging) that is associated with a fall in hemoglobin concentration of 3 to <5 g/dL (or, when hemoglobin concentration is not available, a fall in hematocrit of 9 percent to <15 percent
cardiac death | 12 months
  cardiac death

CONTACTS AND LOCATIONS:
Overall Officials: Mingyou Zhang, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- Jilin university, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Delewi R, Zijlstra F, Piek JJ. Left ventricular thrombus formation after acute myocardial infarction. Heart. 2012 Dec;98(23):1743-9. doi: 10.1136/heartjnl-2012-301962. No abstract available. PMID 23151669
- [Background] Lattuca B, Bouziri N, Kerneis M, Portal JJ, Zhou J, Hauguel-Moreau M, Mameri A, Zeitouni M, Guedeney P, Hammoudi N, Isnard R, Pousset F, Collet JP, Vicaut E, Montalescot G, Silvain J; ACTION Study Group. Antithrombotic Therapy for Patients With Left Ventricular Mural Thrombus. J Am Coll Cardiol. 2020 Apr 14;75(14):1676-1685. doi: 10.1016/j.jacc.2020.01.057. PMID 32273033
- [Background] Kontny F, Dale J, Hegrenaes L, Lem P, Soberg T, Morstol T. Left ventricular thrombosis and arterial embolism after thrombolysis in acute anterior myocardial infarction: predictors and effects of adjunctive antithrombotic therapy. Eur Heart J. 1993 Nov;14(11):1489-92. doi: 10.1093/eurheartj/14.11.1489. PMID 8299630
- [Background] Neskovic AN, Marinkovic J, Bojic M, Popovic AD. Predictors of left ventricular thrombus formation and disappearance after anterior wall myocardial infarction. Eur Heart J. 1998 Jun;19(6):908-16. doi: 10.1053/euhj.1998.0871. PMID 9651715
- [Background] Nadareishvili ZG, Choudary Z, Joyner C, Brodie D, Norris JW. Cerebral microembolism in acute myocardial infarction. Stroke. 1999 Dec;30(12):2679-82. doi: 10.1161/01.str.30.12.2679. PMID 10582996